CLINICAL TRIAL: NCT04711733
Title: Supportive Care Needs of Former Child, Adolescent and Young Adult Cancer Patients, and of Their Parents: Evaluation During Long-term Follow-up
Brief Title: Supportive Care Needs of Former Child, AYA Cancer Patients, and of Their Parents: Evaluation During Long-term Follow-up
Acronym: ExPEDAJAC
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Collaborators: University of Paris 5 - Rene Descartes (Other); Institut d'Hématologie et d'Oncologie Pédiatrique (Unknown)
Responsible Party: Sponsor
Other Study IDs: ET20000319
Record Dates: First submitted 2021-01-11; First posted 2021-01-15 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor or Lymphoma
Keywords: Psycho-oncology; Health Psychology; Paediatric oncology; Supportive care; Survivorship; Caregiver; Children; Adolescents and Young Adults
MeSH Terms: conditions — Lymphoma | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Patients 6-14 years old: Individual interview + Self-report questionnaire + long-term follow-up medical consultation + At 1 year : Assessment of prescription's adherence
  Interventions: Other: Interview; Other: Self-report questionnaire; Other: Medical consultation
- Parents of 6-14 years old patients: Individual interview + Self-report questionnaire
  Interventions: Other: Interview; Other: Self-report questionnaire
- Patients 15-25 years old: Individual interview + Self-report questionnaire + long-term follow-up medical consultation + At 1 year : Assessment of prescription's adherence
  Interventions: Other: Interview; Other: Self-report questionnaire; Other: Medical consultation
- Parents of 15-25 years old patients: Individual interview + Self-report questionnaire
  Interventions: Other: Interview; Other: Self-report questionnaire
- Patients > 25 years old: Individual interview + Self-report questionnaire + long-term follow-up medical consultation + At 1 year : Assessment of prescription's adherence
  Interventions: Other: Interview; Other: Self-report questionnaire; Other: Medical consultation
- Parents of > 25 years old patients: Individual interview + Self-report questionnaire
  Interventions: Other: Interview; Other: Self-report questionnaire

INTERVENTIONS:
Other: Interview — The qualitative interview aims to identify the supportive care needs of patients and parents as well as their expectations with regard to a long-term follow-up.
Other: Self-report questionnaire — To assess the quality of life, anxiety/depression of former patients and relatives:
  For child and adolescent patients (less than 15 years old at inclusion):
  * Pediatric Quality of Life Inventory Cancer module
  * Screen for Child Anxiety Related Emotional Disorders Revised
  * Children's Depression Inventory
  For patients over 15 years of age at the time of inclusion and parents:
  * 36-Item Short Form Health Survey
  * Hospital Anxiety and Depression Scale
  To describe and evaluate the offer and use of the network of health professionals who are aware of post-treatment issues: number of consultations, speciality and location of the professionals requested following the long-term follow-up consultation, time between referral and first consultation, evaluation of the geographical accessibility of care around the patient's home.
Other: Medical consultation — To assess adherence to long-term follow-up medical consultation:
  - number of patients summoned/ number of consultations carried out ; reason for refusal of long-term follow-up medical consultation To assess medical complications through clinical data collection
  Groups: Patients 15-25 years old; Patients 6-14 years old; Patients > 25 years old

SUMMARY:
Each year, there are 2100 new cases of cancer in children and adolescents/young adults (AYA) in France. Due to a significant improvement in the effectiveness of therapies, the survival rate of all types of cancer combined after 5 years is 80-85%. This is leading to the emergence of new problems, which require an adaptation of the long-term care of these former patients. Nevertheless, although some medical complications have been widely described and are the subject of recommendations, many questions remain unanswered regarding the real long-term needs of patients and of their main caregivers.

The main objective of this study is to assess not only the specific supportive care needs of former onco-hematology patients treated before the age of 25 years, but also those of their parents up to 6 months after the end of the oncological follow-up, i.e. 3 to 5 years after the diagnosis.

The secondary objectives aim to:

1. Assess adherence to long-term follow-up medical consultation
2. Assess the early complications presented by the patients
3. Assess the quality of life and the anxiety-depression of former patients and their parents
4. Describe and evaluate the offer and use of the network of health professionals aware of the post-treatment issues; assess the referral to the network of health professionals aware of the post-treatment issues.

Depending on the objectives, the methodology used in this study is mixed, qualitative and quantitative. The study will be proposed systematically to all former patients of the hospital department diagnosed before the age of 25 years and at least 6 years of age at the time of inclusion as well as to their parents. A sample of 60 former pediatric patients (20 per age group) and 60-120 parents (ideally 40 per age group) is expected.

At the scientific level, this study will provide a better understanding of the cognitive and emotional processes involved in the long-term follow-up, in particular by identifying the supportive care needs of different participants (former patients and parents) and their experiences and quality of life during the long-term follow-up phase. At the individual level, this pilot study will enable the development of a multiprofessional structure, expert in cancer after-care from the end of the oncological follow-up.

DETAILED DESCRIPTION:
Rational Each year, there are 2100 new cases of cancer in children and adolescents/young adults (AYA) in France. Due to a significant improvement in the effectiveness of therapies, the survival rate of all types of cancer combined after 5 years is 80-85%. This is leading to the emergence of new problems, which require an adaptation of the long-term care of these former patients. Many studies highlight that 60 to 65% of pediatric oncology patients will present medical and/or psychosocial complications in the 20 years following their oncological treatment, with a cumulative incidence of a serious adverse event of 40% 30 years after the cancer diagnosis. Nevertheless, although some medical complications have been widely described and are the subject of recommendations, many questions remain unanswered regarding the real long-term needs of patients and of their main caregivers, in this project their parents. It is therefore necessary to identify the risk factors by determining the expectations and the supportive care needs of patients and their caregivers in the long-term follow-up in order to intervene early and thus reduce the incidence of these later complications.

However, only 30 to 50% of former patients in pediatric oncology-hematology and their family attend a long-term follow-up medical consultation. We hypothesize that this lack of commitment is multifactorial (e.g. unmet supportive care needs, geographical distance from home, lack of information about the importance of long-term follow-up and follow-up structures nearby) and that a precise study of the needs expressed by former patients and their family should lead to an improved attendance at these consultations.

A better understanding of the supportive care needs of these patients and their families, as well as the brakes/obstacles or lers of their compliance with a long-term follow-up, is therefore essential to improve their quality of life, prevent or detect the sequela of therapies and reduce the risk of morbidity/mortality.

Objectives The main objective of this study is to assess not only the specific supportive care needs of former onco-hematology patients treated before the age of 25 years, but also those of their parents up to 6 months after the end of the oncological follow-up, i.e. 3 to 5 years after the diagnosis.

The secondary objectives aim to:

1. Assess adherence to long-term follow-up medical consultation
2. Assess the early complications presented by the patients
3. Assess the quality of life and the anxiety-depression of former patients and their parents
4. Describe and evaluate the offer and use of the network of health professionals aware of the post-treatment issues; assess the referral to the network of health professionals aware of the post-treatment issues.

Methodology Depending on the objectives, the methodology used in this study is mixed, qualitative and quantitative. The study will be proposed systematically to all former patients of the hospital department diagnosed before the age of 25 years and at least 6 years of age at the time of inclusion as well as to their parents. The experiences and the specific needs of each person (patients, mothers and fathers) will be assessed independently. Three independent groups will be formed based on the age of the patient when included in the study. For each group, the parents may or may not be paired with the patients. A sample of 60 former pediatric patients (20 per age group) and 60-120 parents (ideally 40 per age group) is expected.

Expected results At the scientific level, this study will provide a better understanding of the cognitive and emotional processes involved in the long-term follow-up, in particular by identifying the supportive care needs of different participants (former patients and parents) and their experiences and quality of life during the long-term follow-up phase. This first stage will be followed by more powerful studies on the modalities of following-up patients after cancer, in order to add to previously published research on the long-term medical and psychological side effects.

At the individual level, this pilot study will enable the development of a multiprofessional structure, expert in cancer after-care from the end of the oncological follow-up. This support could be initiated early and the link with the local network established quickly. It should reduce the experience of being abandoned presented by former patients and their families. At the family level, studying the needs expressed by parents could lead to a family psychological approach in order to restore the family links impacted by the disease.

At the organizational level, this study should serve as a basis for developing a structure that can carry out tertiary prevention, and thus reduce the costs attributable to long-term side effects (e.g. educational and professional absenteeism, use of treatments, private consultations or even hospitalization).

ELIGIBILITY:
Inclusion Criteria:

* Age of the patient or the parent of a patient aged ≤ 25 years at diagnosis and at least 6 years of age at the time of inclusion
* Patient, or the parent of a patient, previously treated at Institut d'Hématologie et d'Oncologie Pédiatrique /Leon Berard comprehensive cancer centre
* Patient treated for a solid tumor or a lymphoma
* Patient in complete response and having finished his/her standard oncological monitoring between 1 and 6 months ago i.e. 3 to 5 years after the diagnosis
* Patients and parents capable of understanding, reading and writing French
* Patient affiliated to a health insurance plan
* Having been informed of the study and not objecting to it

Exclusion Criteria:

* Cannot be followed-up for medical, social, familial, geographical or psychological reasons, throughout the duration of the study
* Deprived of liberty by a court or administrative decision
* Person who refused to participate or was incapable of objecting in an informed manner

Ages: 6 Years to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will be proposed systematically to all former patients of the hospital department diagnosed before the age of 25 years and at least 6 years of age at the time of inclusion as well as to their parents. The experiences and the specific needs of each person (patients, mothers and fathers) will be assessed independently. Three independent groups will be formed based on the age of the patient when included in the study. For each group, the parents may or may not be paired with the patients. A sample of 60 former pediatric patients (20 per age group) and 60-120 parents (ideally 40 per age group) is expected. This is the number of interviews after which data saturation generally occurs, i.e. no emergence of new themes from one interview to another.
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Qualitative interview | From 1 to 6 months after the standard monitoring consultation
  To identify the supportive care needs of patients and parents as well as their expectations with regard to a long-term follow-up

SECONDARY OUTCOMES:
Quantitative measures to assess adherence to long-term follow-up medical consultation | From 1 to 6 months after the standard monitoring consultation
  Number of patients summoned/ number of consultations carried out ; reason for refusal of long-term follow-up medical consultation
Clinical Case Report Form to assess the early complications presented by the patients | From 1 to 6 months after the standard monitoring consultation
  Clinical data : cardiac/renal/bones/digestive/hepatic/endocrine/dermatological/sexual/pulmonary/nutritional damages, pain, physical activity, addictology, tiredness, psychological follow-up
Scores of quality of life | From 1 to 6 months after the standard monitoring consultation
  For child and adolescent patients (less than 15 years old at inclusion):
  - Pediatric Quality of Life Inventory Cancer module
  For patients over 15 years of age at the time of inclusion and parents:
  - 36-Item Short Form Health Survey
Scores of anxiety-depression | From 1 to 6 months after the standard monitoring consultation
  For child and adolescent patients (less than 15 years old at inclusion):
  * Screen for Child Anxiety Related Emotional Disorders Revised
  * Children's Depression Inventory
  For patients over 15 years of age at the time of inclusion and parents:
  - Hospital Anxiety and Depression Scale
Quantitative measures to describe and evaluate the offer and use of the network of health professionals who are aware of post-treatment issues | One year after the long-term follow-up consultation
  number of consultations, speciality and location of the professionals requested following the long-term follow-up consultation, time between referral and first consultation, evaluation of the geographical accessibility of care around the patient's home

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Léon Bérard - Institut d'Hémato-Oncologie Pediatrique, Lyon, France

IPD SHARING:
Plan to Share IPD: No